CLINICAL TRIAL: NCT06992414
Title: Exploring Creatine Supplementation for Improved Exercise Capacity and Reduced Fatigue in Long COVID-19: A Randomized Controlled Trial
Brief Title: Exploring the Therapeutic Effects of Creatine Supplementation for Long COVID-19
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Keely Shaw, Postdoctoral Associate, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: REB25-0930
Record Dates: First submitted 2025-05-26; First posted 2025-05-28 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Long COVID Fatigue
Keywords: creatine; post-exertional malaise; exercise; nutraceutical
MeSH Terms: conditions — Motor Activity | interventions — Creatine

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 to the treatment or control group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Creatine monohydrate (Experimental): 8 g/day creatine monohydrate
  Interventions: Dietary Supplement: Creatine monohydrate
- Maltodextrin (Placebo Comparator): 8 g/day maltodextrin
  Interventions: Dietary Supplement: Creatine monohydrate

INTERVENTIONS:
Dietary Supplement: Creatine monohydrate — 8 g/day creatine monohydrate powder

SUMMARY:
Individuals living with Long COVID often experiencing a degree of undue fatigue after physical or cognitive exertion secondary to the condition, timed post-exertional malaise 9PEM). This trial aims to explore the efficacy of creatine monohydrate in managing PEM

DETAILED DESCRIPTION:
cognitive dysfunction, and post-exertional malaise are common complaints of those living with Post-COVID Condition (PCC), a sequelae of symptoms that persist beyond acute infection. Similar to other types of post-viral fatigue, the diagnosis and treatment of PCC are challenging due to the lack of a valid biomarker for the condition. Though the etiology of PCC is not well understood, recent research has found reduced skeletal muscle creatine concentration in those with PCC, which may contribute to fatigue. The objective of this study is to determine if eight weeks of creatine monohydrate supplementation (8g/day) improves symptoms of fatigue, cognition, exercise capacity, and PEM in individuals living with PCC.

Participants will complete two cardiopulmonary exercise tests 24-hours apart on a cycle ergometer before and after an eight-week intervention period. Venous blood samples will be collected before and after exercise on both days to assess changes in mitochondrial function. During the intervention, participants will be randomly assigned to supplement with 8g/day of either creatine monohydrate or a control (maltodextrin). Cognition will be indirectly assessed via self-report of cognitive symptom frequency and severity at baseline, mid-intervention (i.e., 4 weeks) and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Experiencing symptoms at least 3 months after a COVID-19 diagnosis confirmed by positive polymerase chain reaction (PCR) test
* Experiencing post-exertional malaise, as per the DePaul Symptom Questionnaire

Exclusion Criteria:

* Allergy or intolerance to creatine monohydrate or maltodextrin
* Supplemented with creatine in the past eight weeks
* orthopaedic injury or condition that would prevent exercise testing
* change in medication related to Long COVID symptom management in the past month.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-07-02 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Oxygen consumption at ventilatory threshold | From enrollment to the end of intervention at 8 weeks
  point of respiratory compensation point (i.e., ventilatory threshold 2) as a percent of maximal oxygen consumption
Heart rate at ventilatory threshold | From enrollment to the end of intervention at 8 weeks
  heart rate (in bpm) at point of ventilatory threshold

SECONDARY OUTCOMES:
Fatigue | From baseline to mid intervention (4 weeks) to the end of the intervention (8 weeks)
  severity assessed using visual analog scale with zero being not present and 100 being the worst imaginable
Brain fog | From baseline to mid intervention (4 weeks) to post intervention (8 weeks)
  severity assessed using visual analog scale with zero being not present and 100 being the worst imaginable

CONTACTS AND LOCATIONS:
Overall Officials: Keely A Shaw, PhD, Principal Investigator — University of Calgary

IPD SHARING:
Plan to Share IPD: Yes
IPD will be provided upon reasonable request to the PI
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be available beginning ~ December 2026 for 5 years
Access Criteria: IPD will be accessible by reasonable request (email) to the PI